CLINICAL TRIAL: NCT05817565
Title: Outcomes of Physical Therapy Program on Respiratory and Phrenic Nerve Functions in Cervical Disc Compression
Brief Title: Physical Therapy on Phrenic Nerve Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Takey Ahmed, Asssociate Professor, Cairo University
Other Study IDs: respiration and phrenic
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Function Test; Phrenic Nerve Irritation; Cervical Disc Lesion
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention group: Patients underwent physical therapy program 3days/week for three months in the form of
  * Heat therapy by using infrared on the cervical region for relaxation of spasmed neck muscles, while the patient in sitting position.
  * While the patient is sitting, the ultrasound was applied on the para spinal muscles of cervical region for controlling pain.
  * Intermittent cervical traction (traction force equal 8% of body weight) was applied with the patient lying supine and the head in neutral position.
  Interventions: Device: Ultrasound (Phyaction 190 I); with a frequency of 3 MHz was used

INTERVENTIONS:
Device: Ultrasound (Phyaction 190 I); with a frequency of 3 MHz was used — Intermittent cervical traction (traction force equal 8% of body weight) was applied with the patient lying supine and the head in neutral position.
  Other Names: Cervical traction (Eltrac 471); for widening of cervical disc space.

SUMMARY:
This study was conducted to investigate the effects of a designed physical therapy program on respiratory function and phrenic nerve activity in cervical disc compression.

DETAILED DESCRIPTION:
Twenty patients from the Spinal Unite represented the sample of the study. Their mean ages were 43 years and they suffering from acute cervical disc compression at the level of cervical 3, 4, 5. Methods: Evaluation was carried out before and after three months of treatment. It included measuring of pulmonary functions (VC, FVC, FEV1, PEF and MVV) by using spirometer, diaphragmatic excursion and thoracic volume via x-ray and conduction velocity and amplitude of phrenic nerve using electromyography. Treatment program included heat application, ultrasound, cervical traction and diaphragmatic breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

* suffered from cervical disc compression for 6-8 months.
* patients examined and referred by physician.

Exclusion Criteria:

* Any cardio pulmonary disorders which may alter pulmonary function.
* They did not receive any physical therapy program prior to their participation in the study.

Ages: 40 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: study was conducted on 20 patients with compression of the cervical disc at the level of 3, 4, and 5. Their mean age was 43 years; mean weight was 75 kg and mean height was 170cm.They suffered from cervical disc compression for 6-8 months.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
pulmonary function test | 4 months
  to measure vital capacity
phrenic nerve amplitude | 4 months
  objective method to detect phrenic nerve function

CONTACTS AND LOCATIONS:
Overall Officials: Maha m El monem, Ass Prof, Study Chair — Cairo University
Locations (1):
- Cairo University, Giza, Ben El Sarayat, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvalho, M. De (2004) Electrodiagnostic assessment of respiratory dysfunction in motor neuron disease, Handbook of Clinical Neurophysiology. Elsevier B.V. doi: 10.1016/S1567-4231(04)04029-8.